CLINICAL TRIAL: NCT06782737
Title: Effect of the Mediterranean Type Diet Versus Standard Diet on Cardiometabolic Indicator in Patients With Obstructive Sleep Apnea
Brief Title: Mediterranean Diet Versus Standard Diet on Candiormetabolic Indicator in Patients With Apnea
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Lubia Velázquez López, Titular Investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-3609-055
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; obesity; cardiometabolic risk; mediterranean diet; nutritional therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Masking Description: Patients in this group will be given a normocaloric diet with the following energy distribution (Protein: 15-20%, Carbohydrate: 50-55%, Fat: 25-30%, Saturated fat: <7%) according to the guidelines for adult OSA patients. The Mifflin-St. Mifflin equation will be applied to determine the energy needs of each patient. To achieve energy requirements and distribution.
  Patients in this group will receive individual nutritional counseling at the beginning of the study on hygienic sleep measures and Mediterranean-type diet adjusted to foods in Mexico that are accessible and inexpensive. Pre-established menus will be calculated with foods that are characteristic of the Mediterranean-type diet, containing fruits, vegetables, whole grains, cereals, white meat content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Mediterranean diet (Experimental): Patients in this group will be given a normocaloric diet with the following energy distribution (Protein: 15-20%, Carbohydrate: 50-55%, Fat: 25-30%, Saturated fat: <7%) according to the guidelines for adult patients with OSA. The Mifflin-St. Mifflin equation will be applied to determine the energy needs of each patient. They will receive individual nutritional counseling at the beginning of the study on hygienic sleep measures and Mediterranean-type diet adjusted to foods in Mexico. Pre-established menus will be calculated with foods that are characteristic of the Mediterranean-type diet, containing fruits, vegetables, whole grains, cereals, white meat content.
  Sample menus: Weekly menus will be designed to guide the indicated meal plan of the patients. The menus to be designed will be of 1200, 1400, 1600, 1800, 1800, 2000 and 2200 calories. Specifications will be given for the promotion of foods with higher complex carbohydrate content, white meats, fruits and vegetables.
  Interventions: Other: Dietetic interventión with mediterranean diet
- Control (No Intervention): Patients in this group will be given a normocaloric diet with the following energy distribution (Protein: 15-20%, Carbohydrate: 50-55%, Fat: 25-30%, Saturated fat: <7%) according to the guidelines for adult patients with OSA.
  The Mifflin-St. Mifflin equation will be applied to determine the energy needs of each patient. To achieve energy needs and distribution, a specific meal plan containing common foods divided into food equivalent groups will be administered to patients. Nutritional counseling will be considered on an individual basis on hygienic sleep measures and type of diet for weight loss according to age, sex, current body weight and present comorbidity. At the beginning of the intervention, a 24-hour food reminder will be made to know their usual diet. They will be given a triptych for adherence to the indicated diet.

INTERVENTIONS:
Other: Dietetic interventión with mediterranean diet — Personalized dietary Mediterranean diet
  Other Names: Mediterranean diet
  Arms: Intervention Mediterranean diet

SUMMARY:
Introduction. Worldwide, obstructive sleep apnea is estimated to affect one in seven individuals. Patients with OSA present chronic low-grade inflammation related to arteriosclerosis. The effect of the Mediterranean diet on metabolic risk indicators is still inconclusive in the OSA population.

Objective: To evaluate the effect of a Mediterranean diet adapted to the Mexican diet, versus standard nutritional treatment, on metabolic risk indicators in patients with obstructive sleep apnea.

Material and methods: Randomized clinical trial in patients with OSA confirmed by polysomnography. Sociodemographic data, pathological and non-pathological history, as well as clinical data will be collected by interview. Patients will be randomly assigned to the group with personalized Mediterranean-type diet adapted to the Mexican diet or standard diet for patients with OSA. At baseline, 6 and 12 months with the patient fasting, glucose levels and lipid profile in venous blood will be measured, as well as carotid artery thickness. Anthropometry and body composition measurements will also be taken, in addition to questionnaires to measure sleep quality, physical exercise and quality of life, as well as to measure dietary adherence with 3-day food records. A descriptive analysis of qualitative variables will be performed with frequencies and percentages; quantitative variables will be presented according to their free or parametric distribution. An X2 will be performed to compare the difference between the proportions of the outcome variables, as well as a Student's t-test or Mann Whitney U test according to their parametric or free distribution. A multivariate analysis will be performed to see the effect of both interventions on the main outcome variables, obesity, dyslipidemia and glycemic control.

DETAILED DESCRIPTION:
Once the inclusion criteria have been confirmed, a detailed explanation of the study will be given, and the responsible investigators will clarify any doubts about the study. The patient will freely agree to participate in the research by signing the informed consent letter.

The following measurements will be taken in all patients:

Sociodemographic and clinical data. A medical interrogation will be made by the research team to collect sociodemographic data, pathological and non-pathological clinical history. The patient will be questioned about his or her age, clinical history with pathological and non-pathological personal history, pharmacological and non-pharmacological treatment.

Blood Pressure Measurement Blood pressure will be measured by the medical team participating in the study, with a calibrated sphygmomanometer, without previous coffee consumption, without having smoked or consumed cola in the last 30 minutes. The patient will be seated in a chair, with his back supported, without crossing his feet.

. Measurement of sleep variables. In the first time consultation of the Sleep Clinic, parameters of AHI and ODI will be taken with the CPAP equipment, which is part of the studies that are routinely performed in patients with obstructive sleep apnea. It lasts 7 to 8 hours.

Polysomnography: We will proceed to the assembly of the channels that make up the polysomnography: electroencephalographic and electro-oculogram derivations, electromyogram of chin and legs, respiratory flow signals thermistor and/or nasal cannula, respiratory effort signals, continuous oxygen monitoring, electrocardiogram, and determination of the patient's body position.

Measurement of biochemical indicators. With the patient fasting for 8 to 10 hours, a blood sample will be taken in venous blood to measure glucose, lipid profile (Cholesterol, Triglycerides, LDH, VLDL). Measurements to be taken at the first consultation, 6 and 12 months.

Anthropometric and body composition measurements The measurement of the anthropometric data will be done by the nutritionists participating in this research, previously standardized.for the measurement of the body composition the InBody equipment will be used, where the percentage of fat, fat mass, lean mass, total liquids will be obtained.

The Epworth Sleepiness Scale, sleep diary, as well as measures and applied sleep changes will be used. The Epworth Sleepiness Scale (ESE) assesses 8 items, each with a 0 to 3 point response, where 0 means no likelihood of nodding off or falling asleep, 1 means slight likelihood of nodding off or falling asleep, 2 moderate likelihood of nodding off or falling asleep, and 3 high likelihood of falling asleep. If the patient scores 1 to 6 it is considered normal sleep, 7 to 8 points average sleepiness, and 9 to 24 points pathological (abnormal) sleepiness.

Apnea-hypopnea index.

This will be obtained through CPAP readings where the level of severity of OSA before and after the intervention will be calculated. It will be classified:

* Mild: apnea-hypopnea index ≥ 5 and < 15 per hour.
* Moderate: apnea-hypopnea index ≥ 15 and ≤ 30 per hour.
* Severe: apnea-hypopnea index > 30 per hour. Measurement of quality of life It will be obtained from the QSQ questionnaire (Quebec Sleep Questionnaire) which has been validated in Hispanic population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Clinical diagnosis of sleep apnea
* Diagnosis of moderate and severe OSA

Exclusion Criteria:

* Anatomical alterations of the nose, oropharynx or maxilla.
* Chronic kidney disease in substantive treatment of renal function
* Decompensated heart failure
* Cancer
* Depression
* Anxiety
* Neurological disease.
* Treatment with benzodiazepines, antidepressants, anxiolytics and hypnotics.
* Refractory Dyslipidemia
* Familial Dyslipidemia
* Surgeries in less than 6 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
glucose | 12 months
  blood glucose level at baseline and at the end of the study
tryglicerides | 12 months
  Blood triglyceride level at baseline and end of study
body mass index | 12 months
  body mass index

SECONDARY OUTCOMES:
Measurement of sleep quality | The baseline and 12 months after the intervention will be evaluated.
  Measurement of sleep quality The Epworth Sleepiness Scale, sleep diary, as well as measures and applied sleep changes will be used. The Epworth Sleepiness Scale (ESE) assesses 8 items, each with a 0 to 3 point response, where 0 means no likelihood of nodding off or falling asleep, 1 means slight likelihood of nodding off or falling asleep, 2 moderate likelihood of nodding off or falling asleep, and 3 means high probability of falling asleep. If the patient obtains a score of 1 to 6 is considered normal sleep, 7 to 8 points average sleepiness, and 9 to 24 points pathological sleepiness (anaesthesia).
  pathological (abnormal) sleepiness. Apnea-hypopnea index.
Measurement of quality of life | The baseline and 12 months after the intervention will be evaluated.
  It will be obtained from the QSQ questionnaire (Quebec Sleep Questionnaire) which has been validated in the Hispanic population.
  in the Hispanic population. It consists of 32 items focused on measuring daily sleepiness: items 7, 16, 20, 27, 31, 32,
  Daytime symptoms: 1, 10, 11, 14, 17, 17, 18, 19, 23, 26, 29. Nighttime symptoms:
  4, 9, 21, 22, 25, 28, 30. Emotions: 5, 6, 8, 15, 24. Social interactions: 2, 3, 12, 13.
  This questionnaire will be applied at baseline and 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lubia Velazquez, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano Del Seguro Social, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Guillen-Riquelme A, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Buela-Casal G, Ruiz JR. Effect of an Interdisciplinary Weight Loss and Lifestyle Intervention on Obstructive Sleep Apnea Severity: The INTERAPNEA Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e228212. doi: 10.1001/jamanetworkopen.2022.8212. PMID 35452108
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230
- [Background] Godos J, Ferri R, Lanza G, Caraci F, Vistorte AOR, Yelamos Torres V, Grosso G, Castellano S. Mediterranean Diet and Sleep Features: A Systematic Review of Current Evidence. Nutrients. 2024 Jan 17;16(2):282. doi: 10.3390/nu16020282. PMID 38257175
- [Result] Liu Y, Wheaton AG, Chapman DP, Cunningham TJ, Lu H, Croft JB. Prevalence of Healthy Sleep Duration among Adults--United States, 2014. MMWR Morb Mortal Wkly Rep. 2016 Feb 19;65(6):137-41. doi: 10.15585/mmwr.mm6506a1. PMID 26890214
- [Result] Powell TA, Mysliwiec V, Brock MS, Morris MJ. OSA and cardiorespiratory fitness: a review. J Clin Sleep Med. 2022 Jan 1;18(1):279-288. doi: 10.5664/jcsm.9628. PMID 34437054
- [Result] Gaines J, Vgontzas AN, Fernandez-Mendoza J, Bixler EO. Obstructive sleep apnea and the metabolic syndrome: The road to clinically-meaningful phenotyping, improved prognosis, and personalized treatment. Sleep Med Rev. 2018 Dec;42:211-219. doi: 10.1016/j.smrv.2018.08.009. Epub 2018 Sep 3. PMID 30279095
- [Result] Valenza MC, Martin Martin L, Gonzalez Jimenez E, Aguilar Cordero MJ, Botella Lopez M, Munoz Casaubon T, Valenza Demet G. [Risk factors for metabolic syndrome in a population with sleep apnea; evaluation in a population of Granada; the Granada study]. Nutr Hosp. 2012 Jul-Aug;27(4):1255-60. doi: 10.3305/nh.2012.27.4.5825. Spanish. PMID 23165570
- [Result] Salman LA, Shulman R, Cohen JB. Obstructive Sleep Apnea, Hypertension, and Cardiovascular Risk: Epidemiology, Pathophysiology, and Management. Curr Cardiol Rep. 2020 Jan 18;22(2):6. doi: 10.1007/s11886-020-1257-y. PMID 31955254